CLINICAL TRIAL: NCT03310125
Title: Colchicine For The Prevention Of Perioperative Atrial Fibrillation In Patients Undergoing Thoracic Surgery (COP-AF)
Acronym: COP-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-001-COPAF
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Myocardial Injury After Non-Cardiac Surgery
Keywords: Atrial Fibrillation; Inflammation; Thoracic Surgery; Randomized; Colchicine; Myocardial Injury
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Participants received over-encapsulated colchicine 0.5 mg tablet orally twice daily for 10 days.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Participants received matching placebo capsules orally twice daily for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Over-encapsulated 0.5mg tablet twice daily
  Arms: Colchicine
Drug: Placebo — Matching placebo capsule twice daily
  Arms: Placebo

SUMMARY:
The prevention of perioperative atrial fibrillation (AF) and myocardial injury after non-cardiac surgery (MINS) has the potential to reduce mortality, stroke, and hospital stays in patients undergoing major thoracic surgery. Data from cardiac surgery patients suggest that prevention of perioperative atrial fibrillation using an anti-inflammatory agent, such as colchicine, is feasible. The COP-AF trial will assess whether the administration of oral colchicine will reduce the incidence of perioperative atrial fibrillation and myocardial injury after non-cardiac surgery in patients undergoing major thoracic surgery.

DETAILED DESCRIPTION:
Perioperative atrial fibrillation (AF) and myocardial injury after noncardiac surgery (MINS) are among the most common serious complications occurring after thoracic surgery. AF is the most common perioperative cardiac arrhythmia. The incidence of perioperative AF in patients undergoing major thoracic surgery ranges from 10% in low-risk patients to as high as 20% in high-risk patients. The course of patients with perioperative AF is frequently complicated by hemodynamic instability, problems with managing anticoagulation in the early postoperative period, prolonged intensive care unit and hospital stays, and increased costs. Patients who develop perioperative AF (POAF) or MINS also have a significantly increased risk of death and stroke.

Colchicine is an inexpensive drug and a highly effective anti-inflammatory agent that holds great potential for preventing POAF and MINS in patients undergoing thoracic surgery. Data from cardiac surgery patients suggest that prevention of POAF using colchicine is feasible, but whether this concept is also applicable to patients undergoing thoracic surgery, where the risk of POAF is lower and underlying mechanisms may be different, is currently unclear. The 'Colchicine for the prevention of perioperative AF' (COP-AF) trial has been designed as a large randomized, double blind, placebo controlled trial to determine whether colchicine, a potent, safe and inexpensive anti-inflammatory drug, lowers the risk of perioperative AF, MINS, and other inflammatory complications in patients undergoing thoracic surgery. The primary objective of this trial is to determine whether a 10-day course of colchicine 0.5mg twice daily reduces the incidence of perioperative AF and MINS within 14 days after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible if they:

1. are undergoing thoracic surgery with general anesthesia;
2. are greater than or equal to 55 years of age at the time of randomization;
3. are expected to require at least an overnight hospital admission after surgery; and
4. provide written informed consent to participate.

Exclusion Criteria:

Patients will be excluded if they:

1. have a prior history of documented atrial fibrillation;
2. are currently taking anti-arrhythmic medication other than β-blockers, calcium channels blockers or digoxin;
3. are undergoing minor thoracic interventions/procedures (i.e., minor chest-wall surgeries, chest tube insertions, or needle pleural/lung biopsies);
4. have a contraindication to colchicine (i.e., allergy to colchicine, myelodysplastic disorders, or an estimated glomerular filtration rate less than 30 mL/min/1.73m);
5. are not expected to take oral medications for greater than 24 hours after surgery (e.g., esophagectomy);
6. are scheduled for lung transplantation;
7. are currently taking non-study colchicine before surgery;
8. have severe hepatic dysfunction;
9. have aplastic anemia;
10. are a woman of childbearing potential who is pregnant, breastfeeding, or not taking effective contraception;
11. took within the last 14 days or are scheduled to take during the first 10 days after surgery clarithromycin, erythromycin, telithromycin, cyclosporine, ketoconazole, or itraconazole;
12. are an HIV patient treated with antiretroviral therapy; or
13. are scheduled for thoracoscopic lung wedge resection only.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3209 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Clinically important perioperative atrial fibrillation/atrial flutter | 14 days of randomization
Myocardial injury after noncardiac surgery | 14 days of randomization

SECONDARY OUTCOMES:
First occurrence of the composite of all-cause mortality, nonfatal myocardial injury after noncardiac surgery, or nonfatal stroke | 14 days of randomization
First occurrence of the composite of all-cause mortality, nonfatal myocardial infarction, or nonfatal stroke | 14 days of randomization
First occurrence of myocardial injury after noncardiac surgery not fulfilling the 4th universal definition of myocardial infarction | 14 days of randomization
First occurrence of myocardial infarction | 14 days of randomization
Time to chest tube removal | 14 days of randomization
Duration of stay in ICU, step-down, and in-hospital | 14 days of randomization

OTHER OUTCOMES:
Sepsis or infection | 14 days of randomization
  Safety outcome
Non-infectious diarrhea | 14 days of randomization
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: David Conen, MD, MPH, Principal Investigator — Population Health Research Institute; PJ Devereaux, MD, PhD, Study Chair — Population Health Research Institute
Locations (44):
- United States (8):
  - Cleveland Clinic Florida, Weston, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Vienna General Hospital, Vienna, Austria
- Belgium (3):
  - CHU Brugmann UVC, Brussels
  - Hôpital Érasme, Brussels
  - Hôpital Civil Marie Curie, Charleroi
- Canada (12):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Victoria General Hospital, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Victoria Hospital, London, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
- Fundación Cardioinfantil y LaCardio, Bogotá, Cundinamarca, Colombia
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Italy (5):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino, Torino
  - Ospedale Santa Maria della Misericordia, Udine
- Malaysia (2):
  - Hospital Serdang, Kajang, Selangor
  - University of Malaya Medical Centre, Kuala Lumpur, Selangor
- Shifa International Hospital, Islamabad, Islamabad, Pakistan
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- Switzerland (2):
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ofori S, Wang MK, Popova E, McIntyre WF, Chan M, Sessler DI, Giulia V, Warwas M, Balasubramanian K, Tandon V, Finley C, Anna GT, Cata J, Srinathan S, Reimer C, McLean S, Trujillo JC, Fleischmann E, Voltolini L, Cruz P, Maziak DE, Gutierrez-Soriano L, Amir M, Bossard M, Wang CY, Devereaux PJ, Conen D; COP-AF investigators. Smoking, Colchicine and Postoperative Outcomes in Thoracic Surgery: Post Hoc Analysis of the COP-AF Randomized Controlled Trial. CJC Open. 2025 Apr 21;7(7):860-870. doi: 10.1016/j.cjco.2025.04.008. eCollection 2025 Jul. PMID 40698308
- [Derived] Conen D, Ke Wang M, Popova E, Chan MTV, Landoni G, Cata JP, Reimer C, McLean SR, Srinathan SK, Reyes JCT, Grande AM, Tallada AG, Sessler DI, Fleischmann E, Kabon B, Voltolini L, Cruz P, Maziak DE, Gutierrez-Soriano L, McIntyre WF, Tandon V, Martinez-Tellez E, Guerra-Londono JJ, DuMerton D, Wong RHL, McGuire AL, Kidane B, Roux DP, Shargall Y, Wells JR, Ofori SN, Vincent J, Xu L, Li Z, Eikelboom JW, Jolly SS, Healey JS, Devereaux PJ; COP-AF Investigators. Effect of colchicine on perioperative atrial fibrillation and myocardial injury after non-cardiac surgery in patients undergoing major thoracic surgery (COP-AF): an international randomised trial. Lancet. 2023 Nov 4;402(10413):1627-1635. doi: 10.1016/S0140-6736(23)01689-6. Epub 2023 Aug 25. PMID 37640035
- [Derived] Garg AX, Cuerden M, Cata J, Chan MTV, Devereaux PJ, Fleischmann E, Grande AM, Kabon B, Landoni G, Maziak DE, McLean S, Parikh C, Popova E, Reimer C, Trujillo Reyes JC, Roshanov P, Sessler DI, Srinathan S, Sontrop JM, Gonzalez Tallada A, Wang MK, Wells JR, Conen D. Effect of Colchicine on the Risk of Perioperative Acute Kidney Injury: Clinical Protocol of a Substudy of the Colchicine for the Prevention of Perioperative Atrial Fibrillation Randomized Clinical Trial. Can J Kidney Health Dis. 2023 Jul 11;10:20543581231185427. doi: 10.1177/20543581231185427. eCollection 2023. PMID 37457622